CLINICAL TRIAL: NCT05790005
Title: The Effect of the Therapeutic Play Applied Before Surgical Dressing on Anxiety and Fear in Children
Brief Title: The Effect of Therapeutic Play Before Dressing on Anxiety and Fear in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Yeliz Ozer, Principal Investigator, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AMU-SBF-YÖ-01
Record Dates: First submitted 2023-02-23; First posted 2023-03-29 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Anxiety; Fear
Keywords: Anxiety; Fear; Hospitalized Child; Dressings; Play; Operation
MeSH Terms: conditions — Anxiety Disorders | interventions — Play Therapy

STUDY DESIGN:
Intervention Model Description: two groups, the Intervention group and the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): A therapeutic play will be played for 20 minutes after the warm-up play for 10 minutes before the first surgical dressing to be applied after the surgery with children in the 7-12 age groups. There will be 46 children in the intervention group.
  Interventions: Other: therapeutic play
- Control group (No Intervention): Therapeutic play will be not played for 20 minutes after the 10-minute warm-up game before the first surgical dressing to be applied after the surgery with children in the 7-12 age group. The routine procedure applied in the service before the dressing process will be applied. There will be 46 children in the control group.

INTERVENTIONS:
Other: therapeutic play — 2 days after the operation, 1 hour before the dressing, a warm-up game will be played with the child in the playroom of the pediatric surgery service, aiming to put the organs prepared by the researcher in their correct places on the picture for the first 10 minutes. Then, the teddy bear, which is given the appearance of an operation area by sewing a zipper on his stomach, will be given to the child and he will be asked to make the first dressing of the teddy bear. therapeutic game, in which the dramatization method is used, will last 20 minutes. During the 30-minute play practice, the child's questions will be answered.
  Arms: Intervention group

SUMMARY:
The goal of this experimental study is to determine the effect of therapeutic play method applied to hospitalized children aged 7-12 before the first surgical dressing attempt, on anxiety and fear. Researcher will compare the study and control groups to see if therapeutic play has an effect on anxiety and fear.

DETAILED DESCRIPTION:
G-Power 3.1.9.4 package program was used for sample size calculation in the study. Children will be assigned to the study and control groups using the www.randomizer.org program with a simple randomization method to ensure homogeneity between the study and control groups. Before dressing, a warm-up play will be played for 10 minutes with the study group, followed by a 20-minute therapeutic game in which the dramatization method will be used. The children in the control group will be subjected to the routine dressing procedure. The data of the research will be collected using the Child and Parent Information Form, Child Anxiety Scale-State Scale and Child Fear Scale.

During the evaluation of the data, the sociodemographic characteristics of the groups participating in the study will be stated as numbers and percentages, and the normal distribution of the anxiety scale and fear scale scores before the play, after the play and after the dressing process in the Intervention and control groups will be determined by looking at the skewness coefficients. The Factorial Anova Test will be used for mixed measurements in order to examine the anxiety and fear changes of the children in the Intervention and control groups before the play, after the play and after the dressing process. In addition, since this test does not measure the different changes between the groups, the Anova Test in Repeated Measurements will be used to compare the anxiety and fear scores of only the Intervention group and only the control group before the play, after the play and after the dressing process. If the data do not have a normal distribution, the Friedman Test, which is a nonparametric test, will be used.

ELIGIBILITY:
Inclusion Criteria:

* Children in the 7-12 age group
* Children who speak and understand Turkish
* Children whose first dressing will be done in the service on the second day after the operation

Exclusion Criteria:

* Children with hearing, vision and speech problems in themselves or their parents
* Children with a mental disorder in themselves or in their parents
* Children who had circumcision surgery (because the primary dressing was removed and crystallin spray was sprayed on the surgical area and the area was left open)
* Children who should not move before dressing (having hypospadias surgery)
* Children still in the intensive care unit at the time of the first surgical dressing
* Children whose dressing had to be changed before the second postoperative day (wetting, bleeding, opening, etc.)
* Children with previous play therapy experience

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2023-04-07 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Child Anxiety Scale-State Scale | two hours before the surgical dressing
  The scale is shaped like a thermometer with 10 horizontal lines and has a score of 0-10, ranging from calm to very nervous. The child will be asked to mark the anxiety he feels at that moment.
Child Anxiety Scale-State Scale | fifteen minutes before the surgical dressing
  The scale is shaped like a thermometer with 10 horizontal lines and has a score of 0-10, ranging from calm to very nervous. The child will be asked to mark the anxiety he feels at that moment.
Child Anxiety Scale-State Scale | immediately after the surgical dressing
  The scale is shaped like a thermometer with 10 horizontal lines and has a score of 0-10, ranging from calm to very nervous. The child will be asked to mark the anxiety he feels at that moment.
Child fear scale | two hours before the surgical dressing
  The scale consists of five facial expressions that differ from neutral to frightened expressions and scores between 0-4. The child will be asked to choose the facial expression that shows how much the dressing to be applied frightens him.
Child fear scale | fifteen minutes before the surgical dressing
  The scale consists of five facial expressions that differ from neutral to frightened expressions and scores between 0-4. The child will be asked to choose the facial expression that shows how much the dressing to be applied frightens him.
Child fear scale | immediately after the surgical dressing
  The scale consists of five facial expressions that differ from neutral to frightened expressions and scores between 0-4. The child will be asked to choose the facial expression that shows how much the dressing to be applied frightens him.

CONTACTS AND LOCATIONS:
Overall Officials: Hüsniye Çalışır, Prof. Dr., Study Director — Aydin Adnan Menderes University
Locations (1):
- Celal Bayar University Hafsa Sultan Hospital, Manisa, Uncubozköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No